CLINICAL TRIAL: NCT01324167
Title: Effects of Gene Polymorphisms on Metabolic Features in Clozapine-treated Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chun-Hsin Chen, Department of Psychiatry, WanFang Hospital
Other Study IDs: 99037
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators would like to know the association of gene polymorphisms and metabolic adversities in clozapine-treated patients with schizophrenia in Taiwan.

DETAILED DESCRIPTION:
The atypical antipsychotics, such as olanzapine, risperidone, quetiapine, and ziprasidone, are effective in treating both the positive and negative symptoms in schizophrenia (Kelleher et al., 2002). However, atypical antipsychotics have been linked to several forms of morbidity, including obesity, hyperlipidemia, and type 2 diabetes mellitus (DM) (Bergman and Ader, 2005; Jin et al., 2004; Melkersson and Dahl, 2004). Compared with the general population, life expectancy in schizophrenic patients is shorter by as much as 20%, attributable to higher rates of suicide, accidental deaths, and natural causes such as cardiovascular disease and DM (Harris and Barraclough, 1998). Several studies have suggested that these metabolic abnormalities may lead to a greater vulnerability to cardiovascular disease and thus may contribute to the excessive mortality among schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled DSM-IV criteria of schizophrenia or schizoaffective disorder
* 18-65 year of age
* receiving clozapine for at least 6 months

Exclusion Criteria:

* diabetes mellitus patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: schizophrenia or schizoaffective disorder patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-05; Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsin Chen, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan